CLINICAL TRIAL: NCT01814813
Title: A Phase II Randomized Trial Comparing the Efficacy of Heat Shock Protein-Peptide Complex-96 (HSPPC-96) (NSC #725085, ALLIANCE IND # 15380) Vaccine Given With Bevacizumab Versus Bevacizumab Alone in the Treatment of Surgically Resectable Recurrent Glioblastoma Multiforme (GBM)
Brief Title: Vaccine Therapy With Bevacizumab Versus Bevacizumab Alone in Treating Patients With Recurrent Glioblastoma Multiforme That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB futility analysis
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A071101; U10CA031946 (NIH); NCI-2013-00444 (Other: Clinical Trial Reporting Program)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Glioblastoma; Recurrent Adult Brain Tumor; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — vitespin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1, HSPPC-96 + concomitant bevacizumab (Experimental): HSPPC-96 0.4mL intradermal on days 1 and 8 of cycles 1 and 2, then on day 1 of each cycle, up to a maximum of 12 doses (10 cycles), plus bevacizumab 10 mg/kg intravenous (IV) on day 1 of each cycle, until progression. HSPPC-96 should be administered at least 60 minutes prior to starting bevacizumab infusion. (1 cycle=14 days)
  Note: If HSPPC-96 treatment has ended but there is no evidence of disease progression, the patient should continue to receive bevacizumab at the specified dose until progression.
  Interventions: Biological: HSPPC-96; Drug: bevacizumab
- Arm 2, HSPPC-96 with bevacizumab at progression (Experimental): HSPPC-96 0.4mL intradermal on days 1 and 8 of cycles 1 and 2, then on day 1 of each cycle, up to a maximum of 12 doses (10 cycles). At progression: bevacizumab 10mg/kg intravenous (IV) on day 1 of each cycle, until further progression. (1 cycle = 14 days)
  NOTE: It is possible that HSPPC-96 vaccination may end prior to evidence of progression. In this instance it is important to wait until there is confirmed evidence of progression before initiating treatment with bevacizumab.
  Upon confirmation of progression the patient should initiate bevacizumab within 7-42 days from the last dose of vaccine.
  Interventions: Biological: HSPPC-96; Drug: bevacizumab
- Arm 3, Bevacizumab (Active Comparator): Bevacizumab 10mg/kg intravenous (IV) on day 1 of each cycle, until progression. (1 cycle = 14 days)
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Biological: HSPPC-96 — intradermal infusion
  Arms: Arm 1, HSPPC-96 + concomitant bevacizumab; Arm 2, HSPPC-96 with bevacizumab at progression
Drug: bevacizumab — intravenous

SUMMARY:
This randomized phase II trial studies how well giving vaccine therapy with or without bevacizumab works in treating patients with recurrent glioblastoma multiforme that can be removed by surgery. Vaccines consisting of heat shock protein-peptide complexes made from a person's own tumor tissue may help the body build an effective immune response to kill tumor cells that may remain after surgery. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them. It is not yet known whether giving vaccine therapy is more effective with or without bevacizumab in treating glioblastoma multiforme.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects of a vaccine with bevacizumab versus bevacizumab alone on a patient's brain tumor. The vaccine is called heat shock protein peptide complex 96 (HSPPC-96). HSPPC-96 is experimental. Specifically, HSPPC-96 is a protein that may work to help the body have a response against remaining brain tumor cells. Bevacizumab has been approved by the Food and Drug administration for treating brain tumors that grow back. In this study, patients will either get HSPPC-96 vaccine at the same time as bevacizumab, HSPPC vaccine first and then bevacizumab if the tumor comes back, or bevacizumab alone. The use of HSPPC-96 and bevacizumab is investigational.

The primary objective of the study is to determine whether there is an overall survival advantage of HSPPC-96 administered with bevacizumab, given concomitantly or at the point of progression, in comparison with bevacizumab alone in patients with surgically resectable recurrent glioblastoma multiforme.

The secondary objectives are:

1. to evaluate the safety and tolerability of HSPPC-96 with bevacizumab
2. to evaluate the progression free survival of HSPPC-96 with bevacizumab, given concomitantly or at the point of progression.

Patients must undergo surgery within 28 days from pre-registration. There must be confirmation of adequacy of tissue for vaccine manufacture, tumor tissue submitted to Agenus, confirmation of ≥ 90% resection by central radiology review and vaccine manufacture of at least six vials. Patients will be randomized to one of three treatment arms. Please see the "Arms" section for more details.

Patients will be monitored approximately 5 years post-surgery.

ELIGIBILITY:
Pre-registration (Pre-Surgery) Eligibility Criteria

* Histologic documentation: Prior histologic diagnosis of GBM at first occurrence
* Stage: First or second recurrence of GBM or gliosarcoma considered to be surgically resectable
* Prior Treatment:

  * No radiotherapy within 90 days prior to pre-registration
  * No prior treatment with any anti-angiogenic agent targeting the VEGF pathway including but not limited to bevacizumab, cediranib, vandetanib, sunitinib, pazopanib, aflibercept, or sorafenib
  * No prior treatment with HSPPC-96 or other investigational immunotherapy
  * Must have received prior treatment with radiotherapy and temozolomide for histologically confirmed GBM at initial diagnosis
  * No tumor directed therapy for most recent progression
  * No prior Gliadel® wafers
* No clinically significant cardiovascular disease:

  * Patients with a history of hypertension must be well controlled (<150/90) on a regimen of antihypertensive therapy.
  * History of arterial thrombotic events within the past 6 months, including transient ischemic attack (TIA), cerebrovascular accident (CVA), peripheral arterial thrombus, unstable angina or angina requiring surgical or medial intervention in the past 6 months, or myocardial infarction (MI). Patients with clinically significant peripheral artery disease (i.e., claudication on less than one block), significant vascular disease (i.e., aortic aneurysm, history of aortic dissection) are not eligible.
  * Patients who have had a deep vein thrombosis or pulmonary embolus within the past 6 months are eligible if they are on stable therapeutic anticoagulation
  * No current New York Heart Association classification II, III or IV congestive heart failure
* No significant bleeding within the past 6 months; no bleeding diathesis or coagulopathy
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within past 12 months
* No evidence of any systemic autoimmune disease (e.g. Hashimoto's thyroiditis) and/or any history of primary or secondary immunodeficiency, and no immunosuppressant therapy (with the exception of dexamethasone as noted below) for any reason
* Age ≥ 18 years of age
* Karnofsky functional status rating ≥70
* No more than 16 mg dexamethasone (or equivalent) per day
* Non-pregnant and non-nursing

Registration (Post-Surgery) Eligibility Criteria

* Pre-registration eligibility criteria continue to be met
* Histologic documentation: confirmed histological diagnosis of recurrent GBM or gliosarcoma
* ≥ 90% surgical resection of recurrent GBM confirmed by central radiology review by MRI with or without gadolinium per institutional guidelines. A CT scan is allowable in place of MRI only in situations where an MRI is contraindicated (e.g., patient has a heart pacemaker, metallic devices in the eye, brain or spine, severe claustrophobia).
* ≥ 7 grams of resected tumor available for vaccine manufacture as determined by institutional pathologist
* Availability of ≥ 6 clinical vials of HSPPC-96
* Required Initial Laboratory Values:

  * Granulocytes ≥1,500/µL
  * Platelet count ≥100,000/µL
  * Total Bilirubin ≤ 2.0 x ULN
  * UPC ratio <1 or Urine protein ≤ 1+
  * Calculated creatinine clearance ≥ 45 ml/min
  * SGOT/SGPT(AST/ALT) ≤ 2.5 x ULN
* No serious, non-healing wounds or ulcers
* At least 7 days since any minor surgery such as port placement
* No major surgical procedures, open biopsy or significant traumatic injury ≤ 28 days prior to registration or anticipation of need for elective or planned major surgical procedure during the study. Core biopsy or other minor surgical procedures ≤7 days prior to registration.
* No active or recent hemoptysis (≥½ teaspoon of bright red blood per episode) ≤ 30 days prior to registration
* No new bleeding on D28 (+/-3) MRI (or CT if MRI is contraindicated)
* No clinical deterioration at the time of registration/randomization
* If a second surgery is needed for completion of resection, this should be within 30 days from the first surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2023-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Parney, MD, PhD, Study Chair — Mayo Clinic; Orin Bloch, MD, Study Chair — Northwestern University
Locations (417):
- United States (417):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mercy Cancer Center-Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente, Fresno, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Marquette General Hematology Oncology, Marquette, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hemotology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University Pointe, West Chester, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1, HSPPC-96 + Concomitant Bevacizumab: HSPPC-96 0.4mL intradermal on days 1 and 8 of cycles 1 and 2, then on day 1 of each cycle, up to a maximum of 12 doses (10 cycles), plus bevacizumab 10 mg/kg intravenous (IV) on day 1 of each cycle, until progression. HSPPC-96 should be administered at least 60 minutes prior to starting bevacizumab infusion. (1 cycle=14 days) Note: If HSPPC-96 treatment has ended but there is no evidence of disease progression, the patient should continue to receive bevacizumab at the specified dose until progression. HSPPC-96: intradermal infusion bevacizumab: intravenous
- Arm 2, HSPPC-96 With Bevacizumab at Progression: HSPPC-96 0.4mL intradermal on days 1 and 8 of cycles 1 and 2, then on day 1 of each cycle, up to a maximum of 12 doses (10 cycles). At progression: bevacizumab 10mg/kg intravenous (IV) on day 1 of each cycle, until further progression. (1 cycle = 14 days)>
  > NOTE: It is possible that HSPPC-96 vaccination may end prior to evidence of progression. In this instance it is important to wait until there is confirmed evidence of progression before initiating treatment with bevacizumab. Upon confirmation of progression the patient should initiate bevacizumab within 7-42 days from the last dose of vaccine. HSPPC-96: intradermal infusion. bevacizumab: intravenous
- Arm 3, Bevacizumab: Bevacizumab 10mg/kg intravenous (IV) on day 1 of each cycle, until progression. (1 cycle = 14 days) bevacizumab: intravenous
Period: Overall Study
Arm/Group | Arm 1, HSPPC-96 + Concomitant Bevacizumab | Arm 2, HSPPC-96 With Bevacizumab at Progression | Arm 3, Bevacizumab
Started | 29 | 30 | 31
Completed | 29 | 30 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2, HSPPC-96 With Bevacizumab at Progression: HSPPC-96 0.4mL intradermal on days 1 and 8 of cycles 1 and 2, then on day 1 of each cycle, up to a maximum of 12 doses (10 cycles). At progression: bevacizumab 10mg/kg intravenous (IV) on day 1 of each cycle, until further progression. (1 cycle = 14 days) NOTE: It is possible that HSPPC-96 vaccination may end prior to evidence of progression. In this instance it is important to wait until there is confirmed evidence of progression before initiating treatment with bevacizumab. Upon confirmation of progression the patient should initiate bevacizumab within 7-42 days from the last dose of vaccine. HSPPC-96: intradermal infusion. bevacizumab: intravenous
- Total: Total of all reporting groups
Arm/Group | Arm 1, HSPPC-96 + Concomitant Bevacizumab | Arm 2, HSPPC-96 With Bevacizumab at Progression | Arm 3, Bevacizumab | Total
Number analyzed (Participants) | 29 | 30 | 31 | 90
Age, Customized [Count of Participants; unit: Participants]
  <55 | 13 | 12 | 14 | 39
  >=55 | 16 | 18 | 17 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 14 | 25
  Male | 23 | 25 | 17 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 28 | 26 | 26 | 80
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 4
Karnofsky PS [Count of Participants; unit: Participants] — The Karnofsky Performance Scale (PS) Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses.100: Normal no complaints; no evidence of disease.> 90: Able to carry on normal activity; minor signs or symptoms of disease.80: Normal activity with effort; some signs or symptoms of disease.70: Cares for self; unable to carry on normal activity or to do active work.
  Participants
    70 | 6 | 7 | 6 | 19
    80-100 | 23 | 23 | 25 | 71

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The primary endpoint is overall survival (OS), which is defined as the date from study> registration to the date of death, due to any cause.
Time Frame: Up to 5 years post-surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1, HSPPC-96 + Concomitant Bevacizumab | Arm 2, HSPPC-96 With Bevacizumab at Progression | Arm 3, Bevacizumab
Number analyzed (Participants) | 29 | 30 | 31
months | 6.6 [5.4 to 10.4] | 9.2 [5.7 to 11.6] | 10.7 [8.8 to 17.2]
Statistical Analysis 1: Comparison: Arm 1, HSPPC-96 + Concomitant Bevacizumab vs Arm 2, HSPPC-96 With Bevacizumab at Progression vs Arm 3, Bevacizumab; Test type: Superiority; p = 0.16, Log Rank

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time to progression free survival: which is defined as the date from study registration to the date of first observation of disease progression or death due to any cause (whichever comes first). Progressive disease is defined as one or more of the following:New contrast-enhancing lesion outside of radiation field on decreasing, stable, or increasing doses of corticosteroids, increase by > 50% enhancement from the first post-surgical scan, or a subsequent scan with smaller tumor size, and the scan 8 weeks or later on stable or increasing doses of corticosteroids, clinical deterioration not attributable to concurrent medication or comorbid conditions is sufficient to declare progression on current treatment, for patients receiving bevacizumab therapy, significant increase in T2/FLAIR non-enhancing lesion.
Time Frame: Up to 5 years post-surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1, HSPPC-96 + Concomitant Bevacizumab | Arm 2, HSPPC-96 With Bevacizumab at Progression | Arm 3, Bevacizumab
Number analyzed (Participants) | 29 | 30 | 31
months | 3.7 [2.9 to 5.4] | 2.5 [2.0 to 3.5] | 5.3 [3.7 to 8.0]
Statistical Analysis 1: Comparison: Arm 1, HSPPC-96 + Concomitant Bevacizumab vs Arm 2, HSPPC-96 With Bevacizumab at Progression; Test type: Superiority; p < 0.01, Log Rank

3. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 3 years
Population: Patients who started at least one cycle of treatment and were assessed for adverse events were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1, HSPPC-96 + Concomitant Bevacizumab | Arm 2, HSPPC-96 With Bevacizumab at Progression | Arm 3, Bevacizumab
Number analyzed (Participants) | 25 | 28 | 20
Participants
  Grade 3 | 4 | 3 | 5
  Grade 4/5 | 1 | 2 | 1
Statistical Analysis 1: Comparison: Arm 1, HSPPC-96 + Concomitant Bevacizumab vs Arm 2, HSPPC-96 With Bevacizumab at Progression vs Arm 3, Bevacizumab; Test type: Superiority; p = 0.56, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each cycle for patients randomized to the treatment arm; Up to 5 years.
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for patients who completed at least 1 cycle of tx & AEs were assessed. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Arm 1, HSPPC-96 + Concomitant Bevacizumab | Arm 2, HSPPC-96 With Bevacizumab at Progression | Arm 3, Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/25 | 2/28 | 1/20
Serious Adverse Events (participants affected / at risk) | 6/25 | 10/28 | 4/20
Other Adverse Events (participants affected / at risk) | 20/25 | 23/28 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, HSPPC-96 + Concomitant Bevacizumab (N=25) | Arm 2, HSPPC-96 With Bevacizumab at Progression (N=28) | Arm 3, Bevacizumab (N=20)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, HSPPC-96 + Concomitant Bevacizumab (N=25) | Arm 2, HSPPC-96 With Bevacizumab at Progression (N=28) | Arm 3, Bevacizumab (N=20)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (6) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (3)
Blurred vision (Eye disorders) | 2 (9) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 1 (8) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (3)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (7) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (9) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (6) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 1 (14) | 4 (21)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6) | 1 (2) | 4 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (6) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (35) | 8 (27) | 6 (40)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (8) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 1 (1) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 4 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (5) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (7) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (13) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (6) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (3)
Creatinine increased (Investigations) | 0 (0) | 1 (2) | 2 (14)
Lymphocyte count decreased (Investigations) | 6 (16) | 2 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (6) | 1 (1)
Platelet count decreased (Investigations) | 3 (3) | 4 (8) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (7) | 1 (1)
Weight loss (Investigations) | 2 (5) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 3 (5) | 2 (6) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 3 (8) | 3 (4) | 1 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (5) | 2 (6) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 4 (17) | 2 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (15) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (14) | 2 (13) | 1 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (5) | 1 (1) | 2 (4)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (8) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (9) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (11) | 0 (0)
Headache (Nervous system disorders) | 6 (13) | 4 (11) | 5 (7)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (7) | 4 (9) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (11) | 2 (8) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 3 (8) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (3)
Confusion (Psychiatric disorders) | 0 (0) | 2 (15) | 0 (0)
Depression (Psychiatric disorders) | 2 (6) | 1 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (10) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 2 (8) | 8 (38)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (6) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5) | 1 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (10)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Social circumstances - Other, specify (Social circumstances) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 13 (85) | 12 (50) | 13 (75)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (8) | 3 (5) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT01814813/Prot_SAP_000.pdf